CLINICAL TRIAL: NCT01764737
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study Of The Safety, Tolerability, And Pharmacokinetics Of Intravenous VX15/2503 In Patients With Multiple Sclerosis
Brief Title: Evaluation of Safety, Tolerability, and PK of VX15/2503 In Patients With MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15/2503-N-101
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: VX15/2503; Semaphorin 4D; SEMA4D; CD100; safety; tolerability; pharmacokinetics; immunogenicity; multiple sclerosis; monoclonal antibody
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX15/2503 (Experimental)
  Interventions: Drug: VX15/2503
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX15/2503 — single dose intravenous administration
  Arms: VX15/2503
Drug: Placebo — single dose intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of IV administration of VX15/2503 in patients with multiple sclerosis. The escalation part of the study will determine the maximum tolerated dose (MTD) or the Maximum Administered Dose if no MTD is found.

DETAILED DESCRIPTION:
VX15/2503-N-101 is a single ascending dose-escalation, randomized, double-blinded, placebo-controlled study to evaluate the safety and tolerability of IV-administered VX15/2503 in patients with multiple sclerosis. This will be accomplished by using a dose escalation procedure starting at a low dose of VX15/2503 and will continue based on predefined parameters until the maximum tolerated dose is identified. Patients will be randomized at a 4:1 ratio to receive VX15/2503 to placebo. The patients and the study team will be blinded to the treatment that each patient receives.

The study drug, VX15/2503, is a humanized monoclonal antibody that binds to the semaphorin 4D (SEMA4D; CD100) antigen. Experimental evidence suggest that antibody neutralization of SEMA4D may represent a new therapeutic strategy for treating multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-60 years of age who have been diagnosed with MS for at least 1 year as defined by the 2010 revisions to the McDonald criteria
* Has an EDSS score of 0 to 6.5 inclusive at screening
* Has a body mass index of 18 to 32 kg/m2
* Is willing to undergo and has no contraindications to brain MRI
* Willing to use a medically acceptable method of contraception throughout the study period and for 6 months after the dose of VX15/2503, unless patient is surgically sterile or postmenopausal. Women of childbearing potential must have started using adequate contraception at least 2 months before the Day 1 visit.
* Male patients must agree to defer from donating sperm for 6 months after VX15/2503 administration
* Women of childbearing potential must have a negative serum pregnancy test at screening, which will be confirmed at baseline using a urine test before administration of VX15/2503
* Is willing to forego other forms of experimental treatment during the study

Exclusion Criteria:

* Had an MS relapse that did not stabilize within the 30 days before the start of screening.
* Has any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic/gynecologic, pulmonary, neurologic, psychiatric, or renal conditions; has a history of relevant clinically significant allergic or anaphylactic reactions; or has any other clinically significant major disease that, as assessed by the investigator, would pose a risk to patient safety or interfere with the study evaluations, procedures, or completion
* Has any clinically significant laboratory value outside the normal range for MS patients at screening, or has abnormal hematologic, renal, or hepatic function based on laboratory tests
* Is a pregnant or breastfeeding woman
* Has received treatment with any MS disease-modifying therapy other than interferon beta or glatiramer acetate within 3 months prior to dosing
* Has been treated with natalizumab, daclizumab, or fingolimod for any indication within 6 months prior to dosing
* Has had any prior treatment with alemtuzumab, rituximab, mitoxantrone, total lymphoid irradiation, bone marrow transplantation, or T cell or T cell receptor vaccination
* Has received any experimental agent within 6 months prior to dosing, or within a period equivalent to 5 half-lives of the agent (whichever is longer); or is currently involved in any other research study
* Has undergone any major surgical procedure within the 4 weeks prior to dosing
* Has a history of congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to dosing
* Has a clinically significant ECG finding at screening
* Has a known or suspected human immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Has a known or suspected allergy to Gd or other contraindication to brain MRI
* Has a history of an opportunistic infection or a history of acute infection requiring systemic antibiotics, antivirals, or antifungals within 6 weeks prior to dosing (antiinfective therapy must have been completed at least 4 weeks prior to dosing)
* Has any other intercurrent illness or condition, including alcohol or drug dependence as determined by the investigator, which could impact the patient's compliance with or ability to complete the study
* History of seizure disorder or unexplained blackouts or history of seizure within 3 months of screening
* History of suicidal ideation within 3 months prior to screening, episode of severe depression within 3 months prior to screening
* Has a sensitivity to VX15/2503 or the ingredients or excipients of VX15/2503, or known or suspected sensitivity to mammalian cell-derived products
* Has donated or lost more than 1 unit of blood in the 60 days prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability as determined by number of patients with adverse events | Up to 12 weeks depending on dose cohort

SECONDARY OUTCOMES:
Half-life of VX15/2503 | Up to 12 weeks depending on dose cohort
Peak plasma concentration (Cmax) of VX15/2503 | Up to 12 weeks depending on dose cohort
Area under the plasma concentration versus time curve (AUC) of VX15/2503 | Up to 12 weeks depending on dose cohort
Number of patients who develop anti-drug antibody | Up to 12 weeks depending on dose cohort

OTHER OUTCOMES:
Cellular Semaphorin 4D (SEMA4D; CD100) percent saturation | Up to 12 weeks depending on dose cohort
VX15/2503 dose level vs serum SEMA4D levels | Up to 12 weeks depending on dose cohort
Change in magnetic resonance imaging (MRI) parameters as compared to VX15/2503 dose level | Screening to 4 weeks post-dose
  MRI parameters:
  * Number of T1 gadolinium (Gd)-enhancing lesions
  * Number of T2 lesions
  * Total volume of T1 and T2 lesions if the investigational site has the imaging processing capability
VX15/2503 dose vs the change in Kurtzke Expanded Disability Status Scale | Up to 12 weeks depending on dose cohort

CONTACTS AND LOCATIONS:
Overall Officials: John Leonard, PhD, Study Director — Vaccinex Inc.; Keith R Edwards, MD, FAAD, Principal Investigator — MS Center of Northeastern NY/Empire Neurology; Christopher C LaGanke, MD, Principal Investigator — North Central Neurology Associates, PC; T H Rao, MD, Principal Investigator — The Neurological Institute, PA; Lawrence M Samkoff, MD, Principal Investigator — University of Rochester; Lael A Stone, MD, Principal Investigator — The Cleveland Clinic; Omar Khan, MD, Principal Investigator — Wayne State University - University Health Center; Sharon Lynch, MD, Principal Investigator — University of Kansas Medical Center; David H Mattson, MD, Principal Investigator — Indiana University Health Neuroscience Center; Timothy Vollmer, MD, Principal Investigator — University of Colorado Hospital, Anschutz Inpatient Pavilion; Pavle Repovic, MD, Principal Investigator — Swedish Medical Center
Locations (10):
- United States (10):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - University of Colorado Hospital, Aschutz Inpatient Pavilion, Aurora, Colorado
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wayne State University - University Health Center, Detroit, Michigan
  - MS Center of Northeastern NY/Empire Neurology, Latham, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Neurological Institute, PA, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] LaGanke C, Samkoff L, Edwards K, Jung Henson L, Repovic P, Lynch S, Stone L, Mattson D, Galluzzi A, Fisher TL, Reilly C, Winter LA, Leonard JE, Zauderer M. Safety/tolerability of the anti-semaphorin 4D Antibody VX15/2503 in a randomized phase 1 trial. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 16;4(4):e367. doi: 10.1212/NXI.0000000000000367. eCollection 2017 Jul. PMID 28642891
- [Derived] Worzfeld T, Offermanns S. Semaphorins and plexins as therapeutic targets. Nat Rev Drug Discov. 2014 Aug;13(8):603-21. doi: 10.1038/nrd4337. PMID 25082288